CLINICAL TRIAL: NCT04782232
Title: Registry to Assess the Safety and Feasibility of the Subpulmonary Support with the Novel Venous Cannula in Patients with Failing/Absence of the Right Heart
Acronym: RegiVe
Status: Recruiting | Type: Observational
Sponsor: Berlin Heart GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: E-20-325
Record Dates: First submitted 2021-02-15; First posted 2021-03-04 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Univentricular Heart; Ventricular Dysfunction; Heart Diseases; Cardiovascular Diseases
Keywords: EXCOR Ventricular Assist Device; EXCOR Venous Cannula; Failing Fontan
MeSH Terms: conditions — Heart Failure; Univentricular Heart; Ventricular Dysfunction; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with failing/absence of the right heart: Patients with acute or chronic, conservatively uncontrollable heart failure of varying pathogenesis, graded as stage III or IV according to NYHA, with an anticipated need for short-term to long-term right ventricular or biventricular support.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention due to observational design

SUMMARY:
The purpose of the study is to monitor the clinical safety and performance of the EXCOR Venous Cannula in context of an EXCOR VAD therapy to ensure continued acceptability of identified risks, to enable detecting emerging risks and to assess clinical improvement on both short- and long-term.

DETAILED DESCRIPTION:
The registry study has an observational, prospective, international, multi-center, non-randomized design.

The registry is planned for 42 months (3.5 years), with an enrollment period of 28 months, the follow-up of up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient or his/her parent/guardian or legally authorized representative has given the consent by means of a written, signed and dated informed consent form,
* The indications on RVAD and BVAD use of the EXCOR VAD apply,
* Patient shall be on transplant list or at least eligible for HTx,
* BSA (body surface area) greater than or equal to 1.2 m².

Exclusion Criteria:

* Patient or his/her parents/legal guardian or legally authorized guardian has not given the consent,
* The contraindications of EXCOR VAD apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Twenty patients with failing/absence of the right heart. The indications on RVAD and BVAD use of the EXCOR VAD apply.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rate of mortality | 30 days
  Short-term mortality
Rate of major bleeding | 30 days
  Short-term rate of major bleeding
Rate of thrombosis | 30 days
  Short-term rate of thrombosis
Survival to heart transplantation | up to 12 months
  Long-term survival to heart transplantation

SECONDARY OUTCOMES:
Rate of adverse events | up to 12 months
  Safety of the device

CONTACTS AND LOCATIONS:
Locations (1):
- LMU Klinikum, Munich, Germany

REFERENCES:
- [Derived] Dal Sasso E, Schondorf T, Schluter KJ, Miera O, De Rita F, Menon AK; European EXCOR(R) Pediatric Investigator Group (EEPIG). A Novel Strategy for the Mechanical Subpulmonary Support in Failing Fontan Patients. Thorac Cardiovasc Surg. 2022 Dec;70(S 03):e34-e41. doi: 10.1055/s-0042-1757916. Epub 2022 Nov 11. PMID 36368697